CLINICAL TRIAL: NCT07035743
Title: Bronchial Response to Exercise After Double Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: 202500344B0
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Airway Response; Lung Transplant Recipients; Lung Transplant; Challenge Test
Keywords: airway response; double lung transplantation; exercise challenge test; dyspnea; breathlessness
MeSH Terms: conditions — Dyspnea | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- double lung transplant recipients
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 5 minutes of constant workload exercise at 60% of peak oxygen uptake from cardiopulmonary exercise testing
  Other Names: 5-minute exercise
Other: Exercise — 15 minutes of constant workload exercise at 60% of peak oxygen uptake from cardiopulmonary exercise testing
  Other Names: 15-minute exercise

SUMMARY:
This study aims to investigate the airway response to exercise and its association with breathlessness in double lung transplant recipients by comparing responses during 5-minute and 15-minute exercise durations.

DETAILED DESCRIPTION:
Participants will undergo a constant workload challenge set at 60% of their peak oxygen uptake in 2 separate sessions: a 5-minute and a 15-minute exercise session, conducted in a random order. Ratings of perceived exertion will be measured every 5 minutes during exercise. Forced expiratory volume in 1 second will be performed before exercise, immediately post-exercise, and at 5, 10, 15, 20, and 30 minutes post-exercise in order to assess the airway response.

ELIGIBILITY:
Inclusion Criteria:

1. Received double lung transplantation
2. ≥ 3 months post-transplant

Exclusion Criteria:

1. Diagnosis of asthma
2. Significant airflow limitation (≤50% FEV1 predicted)
3. Inability to cooperate with the required tests and measurements
4. Recent infection or rejection within 1 month
5. Exercise contraindication (e.g., recent heart attack or stroke within 3 months, uncontrolled hypertension, known aortic aneurysm, unstable cardiac ischemia, malignant arrhythmias)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: double lung transplantation recipients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in FEV1 from baseline | from enrollment to up to 12 weeks
  Percentage change in FEV1 from baseline at immediately post-exercise, 5, 10, 15, 20, and 30 minutes post-exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zantah M, Pandya A, Marchetti N, Jacobs MR, Criner GJ. Lung Denervation and Its Effect on Bronchial Responsiveness Following Lung Transplant Surgery2020.
- [Background] Stanbrook MB, Kesten S. Bronchial hyperreactivity after lung transplantation predicts early bronchiolitis obliterans. Am J Respir Crit Care Med. 1999 Dec;160(6):2034-9. doi: 10.1164/ajrccm.160.6.9801037. PMID 10588625
- [Background] Reid DW, Walters EH, Johns DP, Ward C, Burns GP, Liakakos P, Williams TJ, Snell GI. Bronchial hyperresponsiveness and the bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2005 Apr;24(4):489-92. doi: 10.1016/j.healun.2004.02.006. PMID 15797754
- [Background] Herve P, Picard N, Le Roy Ladurie M, Silbert D, Cerrina J, Le Roy Ladurie F, Chapelier A, Dartevelle P, Simonneau G, Parquin F, et al. Lack of bronchial hyperresponsiveness to methacholine and to isocapnic dry air hyperventilation in heart/lung and double-lung transplant recipients with normal lung histology. The Paris-Sud Lung Transplant Group. Am Rev Respir Dis. 1992 Jun;145(6):1503-5. doi: 10.1164/ajrccm/145.6.1503. PMID 1596027
- [Background] Glanville AR, Theodore J, Baldwin JC, Robin ED. Bronchial responsiveness after human heart-lung transplantation. Chest. 1990 Jun;97(6):1360-6. doi: 10.1378/chest.97.6.1360. PMID 2140767
- [Background] Glanville AR, Gabb GM, Theodore J, Robin ED. Bronchial responsiveness to exercise after human cardiopulmonary transplantation. Chest. 1989 Aug;96(2):281-6. doi: 10.1378/chest.96.2.281. PMID 2666042